CLINICAL TRIAL: NCT03580785
Title: Primary Failure of Eruption (PFE) : Highlighting of Clinical, Radiological and Genetic Diagnostic Criteria: Consequences on the Therapeutic Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6641
Record Dates: First submitted 2018-04-05; First posted 2018-07-09 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Primary Failure of Eruption
MeSH Terms: interventions — Genetic Testing; Radiography, Panoramic

STUDY DESIGN:
Intervention Model Description: single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: genetic analysis — saliva is collected for DNA extraction
Radiation: panoramic radiography — panoramic radiography
Radiation: teleradiography — teleradiography
Radiation: intraoral X-rays — intraoral X-rays
Radiation: CT scan of maxillary and mandible — CT scan of maxillary and mandible

SUMMARY:
The primary purpose of the study is to identify clinical, radiological and genetic diagnostic criteria for Primary Failure of Eruption (PFE).

The secondary purposes are to highlight the genotype-phenotype correlations in the PTHR1 and non-PTHR1 forms and analyze the therapeutic failures.

ELIGIBILITY:
Inclusion criteria:

* people over 6 years old
* people with Primary Failure Eruption

Exclusion criteria:

* children under 6 years old
* endocrine pathology that may interfere with dental eruption
* rickets
* chemotherapy / radiotherapy
* bisphosphonate treatment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
Number of teeth | at inclusion (day 1)
  number of teeth
Recording of dental caries | at inclusion (day 1)
  recording of dental caries by Decayed Missing Filled Teeth index (DMFT index)
Recording the location of dental caries | at inclusion (day 1)
  the number of teeth affected using the international classification index
Drugs intra uterine exposure | at inclusion (day 1)
  drugs during pregnancy
Nutritional deficiencies | at inclusion (day 1)
  nutritional deficiencies assessed by a questionnaire
Periodontium | at inclusion (day 1)
  assessment of the periodontium by Maynard and Wilson classification
Oral hygiene | at inclusion (day 1)
  assesment of oral hygiene by plaque index (Löe and Silness, 1963)
Gingival inflammation | at inclusion (day 1)
  assesment of gingival inflammation by gingival index (Löe and Silness, 1963)
Treatment needs | at inclusion (day 1)
  assessment of treatment needs using Community Periodontal Index of treatment Needs (CPITN)
Face shape | at inclusion (day 1)
  assesment of the face shape : round, square, oval
Symmetry of the face | at inclusion (day 1)
  symmetry of the face (yes/no)
Profile (shape) | at inclusion (day 1)
  assessment of the profile (shape)
Smile | at inclusion (day 1)
  morphology of the smile
Vertical dimension | at inclusion (day 1)
  assessment of the vertical dimension: anterior infraclusion or overbite (in %)
Transversal dimension | at inclusion (day 1)
  assessment of the transversal dimension: posterior transversal dimension (in mm)
Sagittal dimension | at inclusion (day 1)
  Assessment of the sagittal dimension by Angle's classification
Chewing | at inclusion (day 1)
  Assessment of chewing by Plana's Functional Masticatory Angles (PFMA)
Nasal breathing | at inclusion (day 1)
  Assessment of nasal breathing by the Rosenthal's test
Swallowing | at inclusion (day 1)
  Assessment of swallowing by lingual interposition

SECONDARY OUTCOMES:
Mutations causing PFE | at inclusion (day 1)
Type of treatment performed | at inclusion (day 1)
  (orthodontics, surgery, prothesis)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique dentaire, Strasbourg, France